CLINICAL TRIAL: NCT07209332
Title: An Open-Label Extension Study to Investigate the Long-term Safety, Tolerability, Pharmacokinetics, and Efficacy of WVE-N531 in Patients With Duchenne Muscular Dystrophy Who Participated in Another Study of WVE-N531
Brief Title: Open-Label Extension Study of WVE-N531 in Patients With Duchenne Muscular Dystrophy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVE-N531-002
Record Dates: First submitted 2025-08-14; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- WVE-N531 (Experimental)
  Interventions: Drug: WVE-N531

INTERVENTIONS:
Drug: WVE-N531 — WVE-N531 is an antisense oligonucleotide (ASO)

SUMMARY:
This is a Phase 2 open-label extension (OLE) study to evaluate the long-term safety, tolerability, efficacy, pharmacokinetics, and the pharmacodynamics (PD) through potential exploratory biomarker(s) of intravenous (IV) WVE-N531 in patients with DMD who participated in another study of WVE-N531. All patients will have rolled over from a previous study of WVE-N531.

DETAILED DESCRIPTION:
The study will include up to 175 patients from planned and ongoing WVE-N531 studies globally. All patients will continue to receive 10 mg/kg WVE-N531 IV every 4 weeks (Q4W), through Week 96. Safety monitoring will occur for approximately 11 months after the final dose. The primary objective of the study is to evaluate the long-term safety and tolerability of WVE-N531.

ELIGIBILITY:
Inclusion Criteria:

1. Participated in a prior study of WVE-N531 and has not experienced any significant toxicities due to WVE-N531 or significant clinical deterioration of general health since the last dose or early discontinuation visit.
2. Of note: if there will be a greater than 31-day gap between the last dose on the prior study and the FD on this study, the case should be discussed between the Investigator and Medical Monitor.

Exclusion Criteria:

1. Any clinically significant medical finding or change during or following participation in the prior WVE-N531 study, other than DMD that, in the judgment of the Investigator, would affect the potential safety of the patient to receive WVE-N531 or interfere with participation in the study.
2. Any recreational substance use (including prescribed cannabinoids), with the exception of alcohol and nicotine, irrespective of legality, within 2 months prior to FD and/or unwilling to refrain from such use for the duration of the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by the following parameters: | Time Frame: Week 0 through Week 96
  * Complete Physical examination, including height and weight
  * Vital Signs (via blood pressure, temperature and pulse)
  * Safety Laboratory Tests (including complete blood cell count, urinalysis and clinical chemistry)
  * ECG (12- Lead single tracing)
  * ECHO (including left ventricular ejection fraction)
  * Pulmonary Function Tests (including Peak Flow Rate, Cough Peak Flow, Forced Vital Capacity and Maximum Inspiratory Pressure)

SECONDARY OUTCOMES:
North Star Ambulatory Assessment (NSAA) (Version 2.0) composite score, each item assessed using a 3 point scale, including: | At baseline Week 0 through Week 96
  * Time to stand (measured in seconds )
  * Timed 10-meter walk/run (measured in seconds)
  * Four-stair climb time (measured in time to climb 4 stairs in seconds)
Performance of the Upper Limb (PUL) (Version 2.0) (measured by total score and score of high level shoulder dimension, Mid-level Elbow Dimension, Distal Wrist and Hand Dimension) | At baseline Week 0 through Week 96
Stride Velocity 95th Centile (SV95C) (collected in 3 consecutive weeks) | At baseline Week 0 through Week 96
Upper limb proximal strength (assessed by handheld myometer measured in Kilograms) | At baseline Week 0 through Week 96

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (3):
- Jordan (2):
  - Istiklal Hospital/ Clinical Research Unit, Amman
  - The Specialty Hospital (TSH)/ Advanced Clinical Center, Amman
- Oxford Children's Hospital, Oxford University Hospitals NHS Foundation Trust, Headington, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No